CLINICAL TRIAL: NCT04875923
Title: Cardiac Surgery as a Means of Reversing Frailty - The CURE-Frailty Trial
Brief Title: Cardiac Surgery as a Means of Reversing Frailty
Acronym: CURE-Frailty
Status: Completed | Type: Observational
Sponsor: Dr. Valerie-Anna Rudas (Other)
Responsible Party: Sponsor-Investigator, Dr. Valerie-Anna Rudas, Resident Dept. of Anesthesia, Critical Care and Pain Medicine, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: 1001/2021
Record Dates: First submitted 2021-04-21; First posted 2021-05-06 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Frailty
Keywords: Frailty; Cardiac Surgery
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Frailty is a multifactorial condition associated with older age, which leads to increased vulnerability to external stressors, such as infections or surgical procedures. Key features of frailty are unintentional weight loss, reduced strength and physical activity as well as the feeling of exhaustion.

When selecting patients for surgery, frailty can play an important part in resource planning and prognostication. Multiple studies have shown frailty to have a negative impact on mortality, perioperative adverse events, hospital length of stay as well as postoperative quality of life and functional status. Despite it being an important patient-centered outcome, postoperative quality of life tends to be overlooked when selecting patients for surgery.

Cardiac surgery presents a massive stressor to the frail patient, but on the other hand might have the ability to reduce disease burden and improve functional status, thus reducing frailty.

This prospective observational cohort study aims to assess frailty, as well as functional status and quality of life in cardiosurgical patients pre- and postoperatively, and evaluate its impact on postoperative clinical and functional outcomes.

The primary endpoint of this study is the change in postoperative level of frailty.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 60 years
* elective cardiac surgery

Exclusion Criteria:

* age < 60 years
* emergency procedures
* pulmonary thromboendarterectomy
* declined informed consent
* pregnant women

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing an elective cardiac surgical intervention
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Change in Postoperative Level of Frailty | 12 months
  The "Clinical Frailty Scale" (CFS) will be used to assess frailty. A CFS of 1 indicates absence of frailty, whereas a CFS of 9 indicates severe frailty. A postoperative change in the CFS indicates a postoperative change in frailty.

SECONDARY OUTCOMES:
Quality of Life assessed by the "SF-12 Patient Questionnaire" | 12 months
  Quality of Life will be assessed using the SF-12 Patient Questionnaire.
Functional Status assessed by the "Functional Independence Measure" | 12 months
  Functional status will be assessed using the "Functional Independence Measure", with lower scores indicating a worse functional status.
30-day Mortality | 30 days
  Number of participants who have died within 30 days postoperatively.
Overall Mortality | 12 months
  Number of participants who have died within the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Bernardi, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria